CLINICAL TRIAL: NCT01761864
Title: The Effect of Academic Detailing on Prescribing of Analgesics in Primary Care: a Randomised Controlled Trial
Brief Title: The Effect of Industry-independent Visits to Primary Care Physicians on Medication Prescribing for Pain Relief in Chronic Joint Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Veronique Verhoeven, professor, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: FARMACA007
Record Dates: First submitted 2013-01-02; First posted 2013-01-07 (Estimated); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Study Focus: Prescribing of Drugs

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention group (Experimental): academic detailing receiver
  Interventions: Behavioral: academic detailing intervention
- control group (No Intervention): not receiving an academic detailing intervention

INTERVENTIONS:
Behavioral: academic detailing intervention
  Other Names: academic detailing intervention on evidence-based prescribing of analgetics in chronic joint pain
  Arms: intervention group

SUMMARY:
Osteoarthritis is a common problem in primary care. Long-term use of non-steroidal anti-inflammatory drugs (NSAIDs) for pain relief can lead to serious (gastro-intestinal, cardiovascular and renal) adverse events, that can even result in death. NSAIDs differ in their risk of side effects. Opoid analgesics are sometimes used as an alternative for NSAIDs in patients with osteoarthritis. However, these drugs also can lead to serious adverse events. Simple analgesics are first line treatment in patients with osteoarthritis. NSAIDs and opoid analgesics should be avoided whenever possible.

Farmaka (www.farmaka.be) is a non-profit organisation that operates a nationwide academic detailing service in Belgium since 2006. The academic detailing exists of face-to-face educational visits to general practitioners in their practice by a trained visitor with a medical science degree. The aim of these visits is to improve the quality of drug prescribing in primary care. Small scale experiments in the past showed that academic detailing can indeed improve prescribing behavior.

The current study wants to examine if nationwide academic detailing on appropriate prescribing of analgesics for chronic pain in osteoarthritis results in a better GP's prescribing behavior.

Another research question is whether physician-visitors have more influence on prescribing than non-physician visitors.

It is also interesting to examine if the effect of a visit is larger if there exists a longstanding relationship between the academic detailer and the GP.

About 4.000 general practices are located in a region where academic detailers of Farmaka are operational and have received a visit at least once before. All these practices will be divided into two study groups in a random manner.

The first group of practices will belong to the treatment group. GP's from this group will be offered a face-to-face visit on appropriate prescribing of analgesics for chronic pain in osteoarthritis. The visits will take place between February and June 2013.

The second group of practices will serve as a control group. GP's from these practices won't be offered any visit at all during the year 2013.

Reimbursement data for all GP's are available by request from the Belgian Intermutualistic Agency (IMA). IMA data for 2013 will be available by the end of 2014. These data will allow comparison between the treatment and control group on the amound and type of prescriptions for analgesics in patients with chronic osteoarthritis pain.

A comparison of the prescriptions of practices that participate in the study and the prescriptions of in practices that don't participate is also possible.

The project is funded by the Federal Agency for Medicines and Health Products. We hypothesize that

* the academic detailing visits to GP practices on prescribing of analgesics for chronic pain in osteoarthritis will improve prescribing of analgesics by at least 5%
* the personal relation between the GP and the academic detailer, expressed as the number of previous visits, is an important effect modifier

ELIGIBILITY:
Inclusion Criteria:

* Professionally active GPs of all Belgian primary care practices that have received a visit before by Farmaka and are located in the regions where academic detailers are currently active. No age or gender restrictions.

Exclusion Criteria:

* GPs who are not professionally active (anymore) in a practice located in a region were an academic detailer operates in the period of the visits on analgesics; GP's who have never received an academic detailing visit before.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4000 (Actual)
Dates: Start 2013-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
recommended prescribing of analgetics | 1 year
  Short-term (1 month), intermediate (6 months) and long-term (<= 1 year) use of
  * paracetamol, ibuprofen , naproxen, oxicams, coxibs, nabumeton, tramadol, tilidine;
  * recommended NSAIDs among those treated with NSAIDs expressed as percentage;
  * PPI among those treated with NSAIDs expressed as percentage in insured individuals over 60 years of age and their relevant subgroups.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Antwerp, Wilrijk, Belgium

REFERENCES:
- [Derived] Bruyndonckx R, Verhoeven V, Anthierens S, Cornelis K, Ackaert K, Gielen B, Coenen S. The implementation of academic detailing and its effectiveness on appropriate prescribing of pain relief medication: a real-world cluster randomized trial in Belgian general practices. Implement Sci. 2018 Jan 10;13(1):6. doi: 10.1186/s13012-017-0703-8. PMID 29316945